CLINICAL TRIAL: NCT01501201
Title: Comparison of Gastric By-Pass and Optimized Medical Treatment in Obese Diabetic Patients in Terms of Mortality, Glycemic Control, and Cost Effectiveness - Prospective, Multicenter, Randomized Study
Brief Title: Comparison of Gastric By-Pass and Optimized Medical Treatment in Obese Diabetic Patients
Acronym: DIABSURG
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010_07/1019; 2010-A01141-38. (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2011-12-20; First posted 2011-12-29 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Obesity; Diabetes
Keywords: Obesity; Diabetes; Bariatric Surgery
MeSH Terms: conditions — Obesity; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gastric By-Pass (Experimental): group treated with Gastric By-Pass
  Interventions: Procedure: Gastric By-Pass
- optimized medical management (Active Comparator): group receiving an optimized medical management
  Interventions: Drug: optimized medical management

INTERVENTIONS:
Procedure: Gastric By-Pass — Bariatric surgery laparoscopic Roux-en-Y Gastric Bypass (RYGBP)
  Other Names: RYGBP
  Arms: Gastric By-Pass
Drug: optimized medical management — group receiving an optimized medical management, among patients with obesity and poorly controlled type 2 diabetes
  Arms: optimized medical management

SUMMARY:
The objectives are to compare the results of the Gastric By-Pass (GBP) to that of optimized medical therapy in patients with obesity and poorly controlled type 2 diabetes in terms of mortality, weight loss, glycemic control, quality of life, cost, cost-effectiveness and cost utility of these two strategies.

DETAILED DESCRIPTION:
Optimizing the management of type 2 diabetes (T2D) will remain a major public health concern for decades to come. T2DM has already affected 4% of the French population and generates each year over 12 billion euros of expenditure. By combining therapies, oral and/or injectable (insulin or analogues of GLP-1), the current management of T2DM provides two thirds of patients with a satisfactory metabolic control (HbA1c < 7%) and reduced incidence of cardiovascular complications. Its effect on mortality, however, remains more limited, presumably because of the persistence of other cardiovascular risk factors. A recent study has confirmed that French patients with T2DM present an overall mortality risk significantly higher than the general population. In France, this group registered a mortality of 32 deaths per 1000 persons.

Bariatric surgery is now a recognized method for the treatment of severe obesity. It allows for the permanent loss of at least 50% of initial excess weight. In obese patients, this surgery is also associated with a significant reduction in cardiovascular risk factors and particularly T2D. A recent meta-analysis of retrospective studies available suggests that surgery results in remission of T2DM in over 75% of cases. The only prospective randomized study showed that gastric restriction by placing a gastric band, provides better glycemic control than just medical treatment in obese patients with recently discovered T2DM. The gastric by-pass (GBP) which also includes an intestinal by-pass, seems to have an even higher metabolic efficiency than gastric bypass alone. In patients with T2DM, the GBP restores postprandial insulin secretion independently of weight loss. Despite the significant morbidity of the intervention, long-term results seem broadly supportive of the GBP. In a large case-control study, GBP was associated with a decrease of 90% of deaths related to diabetes. In a controlled study conducted in surgical candidates obese diabetics, the GBP decreased the overall world mortality by 75% after 6 years. Despite these very encouraging data, the GBP is now proposed to only a small proportion (< 1%) of patients likely to benefit from the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus with HbA1c > 7.5 %
* Body mass index > 35 and < 50 kg/m2
* Candidate for Gastric By-Pass
* Treatment with GLP1 (glucagon-like peptide) analogue or insulin

Exclusion Criteria:

* Contraindication to bariatric surgery
* Pregnancy
* Affiliation of health care assurance
* Psychiatric disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 490 (Estimated)
Dates: Start 2011-08-08 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
overall mortality | 5 years
  to compare the results of the GBP to that of optimized medical therapy in patients with obesity and poorly controlled type 2 diabetes in terms of mortality

SECONDARY OUTCOMES:
overall mortality | 7 years
  The objectives are to compare the results of the GBP to that of optimized medical therapy in patients with obesity and poorly controlled type 2 diabetes in terms of mortality
overall mortality | 10 years
  The objectives are to compare the results of the GBP to that of optimized medical therapy in patients with obesity and poorly controlled type 2 diabetes in terms of mortality
weight loss | 2 years
  The objectives are to compare the results of the GBP to that of optimized medical therapy in patients with obesity and poorly controlled type 2 diabetes in terms of weight loss
glycemic control | 2 years
  The objectives are to compare the results of the GBP to that of optimized medical therapy in patients with obesity and poorly controlled type 2 diabetes in terms of glycemic control
quality of life | 2 years
  The objectives are to compare the results of the GBP to that of optimized medical therapy in patients with obesity and poorly controlled type 2 diabetes in terms of quality of life
cost, cost-effectiveness and cost utility | 2 years
  The objectives are to compare the results of the GBP to that of optimized medical therapy in patients with obesity and poorly controlled type 2 diabetes in terms of cost, cost-effectiveness and cost utility of these two strategies.

CONTACTS AND LOCATIONS:
Overall Officials: Francois Pattou, Professor, Study Director — University Hospital of Lille
Locations (10):
- France (10):
  - University Hospital of Lille, Lille, Nord
  - Centre Hospitalier Regional D' Angers, Angers
  - Hopital de Bois-Guillaume Chu Rouen, Bois-Guillaume
  - Hu Ouest Site Ambroise Pare Aphp -, Boulogne-Billancourt
  - Hopital Jeanne D'Arc Chu Nancy, Dommartin-lès-Toul
  - Hopital Lyon Sud - Hcl - Pierre Benite, Lyon
  - Hopital Lapeyronie Chu Montpellier, Montpellier
  - Hu Pitie Salpetriere Aphp, Paris
  - Hopital Larrey Chu Toulouse, Toulouse
  - Ch Valenciennes, Valenciennes

IPD SHARING:
Plan to Share IPD: No